CLINICAL TRIAL: NCT01012986
Title: "Reading Subtitles Skills in the Elementary School"
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Michele Viana Minucci, University of Sao Paulo
Other Study IDs: reading subtitles in Brazil
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Reading Comprehension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 2nd Grade: students of 2nd grade
  Interventions: Other: Assessment of reading skills
- 4th Grade: students of 4th Grade
  Interventions: Other: Assessment of reading skills

INTERVENTIONS:
Other: Assessment of reading skills

SUMMARY:
Theme: The reading of fixed texts in school are widely known, however it is not known how they read texts furniture and what skills are required for this type of reading.

Objective: To evaluate the skills of reading film subtitles in students of 2nd and 4th grade of elementary school of a Public School.

Method: Review the level and skills of reading movies subtitles (RMS), through the recounting of a section of film watched, alone, mute and legend, for 60 students (30 2nd grade and 30 of the 4th grade) matched for age and gender.

DETAILED DESCRIPTION:
The purpose of this study was to compare the reading film subtitles skills in students aged 2nd and 4th grade of elementary school (EF) from a public school, and relate the performance of literacy in school with reading film subtitles.

Proceedings: The study included 30 students from 2nd and 30 from 4th grade of a public school at Sao Paulo. The participants' ages ranged from 7 years and 8 months to 9 years and 3 months in the 2nd grade, and 9 years and 9 months to 11 years and one month in the 4th grade. The groups were matched for the genre.

Inclusion criteria: sign a consent to search, be literate, do not have any sensory changes, and never repeated a grade. Each subject, individually, was rated about the level of literacy and reading through the protocol of school literacy; and about reading film subtitles skills.Each subject recounted what he understood and responded to five inferential questions about the movie.The recount was analyzed and scored on a specific protocol based on Castillo (1999).Students could score in four levels: decoding, literal comprehension, comprehension independent and critical reading.

ELIGIBILITY:
Inclusion Criteria:

* sign a consent to search
* be literate
* do not have any sensory changes
* and never repeated a grade

Ages: 7 Years to 9 Years | Sex: All
Age Groups: Child
Study Population: students in 2nd and 4th grade
Sampling Method: Probability Sample
Enrollment: 60 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - University of Sao Paulo, São Paulo, São Paulo
  - University of São Paulo, São Paulo, São Paulo